CLINICAL TRIAL: NCT00760747
Title: A Randomized, Controlled, Open-Label Comparison Study of the Efficacy and Safety of Slow Transitioning Compared With Fast Transitioning From a Stimulant Medication to Atomoxetine in Pediatric and Adolescent Outpatients With DSM-IV Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Comparison of Slow and Fast Transition From Stimulants to Atomoxetine in Children and Adolescents With Attention Deficit/Hyperactivity Disorder(ADHD)
Acronym: ADHD SWITCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12305; B4Z-EW-LYFJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2011-09-01 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2011-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Children; Stimulant; Atomoxetine; Adolescents
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Slow Switching Group (Experimental): Slow Switching Group (switch from full stimulant dose to atomoxetine, 1.2 mg/kg/day, orally (PO), during 10 weeks then continue treatment up to 1.8 mg/kg/day, PO to 14 weeks
  Interventions: Drug: Atomoxetine
- Fast Switching Group (Experimental): Fast Switching Group (switch from full stimulant dose to atomoxetine 1.2 mg/kg/day, PO, during 2 weeks then continue treatment up to 1.8 mg/kg/day, PO to 14 weeks
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — 1.2 mg/kg/day up to 1.8 mg/kg/day, orally (PO)
  Other Names: LY139603; Strattera

SUMMARY:
Children and adolescents with Attention Deficit Hyperactivity Disorder (ADHD) who are not tolerating or not responding well to stimulant therapy will be included in this study. Two different strategies for transition from Stimulant to Atomoxetine will be used: Slow (10 weeks) and fast (2 weeks). Changes in ADHD symptoms and tolerability of medication will be compared between the two different switching approaches.

DETAILED DESCRIPTION:
Study B4Z-EW-LYFJ is a phase IV multicentre, open label, controlled study in approximately 120 patients with ADHD from 6 years to 16 years of age. After the screening period, patients will be randomized (centrally in a 1:1 ratio) either to a transition period of 10 weeks (slow switching arm) or to a transition period of 2 weeks (fast switching arm). After completion of the 10 week open phase patients will be treated for a further 4 weeks with atomoxetine.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients between 6-16 years of age
* Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) diagnostic criteria for ADHD must be met
* Normal laboratory and electrocardiogram (ECG) results
* Normal intelligence
* Must have unsatisfactory symptom response to stimulant therapy or experience of adverse events while on stimulant therapy

Exclusion Criteria:

* Less than 20 kg or more than 70 kg at study entry
* Concomitant major psychiatry disorders, drug or alcohol abuse or serious suicide risk
* Medical conditions such as seizures, severe allergies, glaucoma, cardiovascular disease, hypertension, or acute or unstable medical conditions
* Taking of anticonvulsants, antihypertensive agents, medication with sympathomimetic activity, psychotropic medications, monoamine oxidase inhibitor
* Immediate need for stimulant discontinuation due to tolerability problems
* Previous participation in an atomoxetine study, or unresponsive to atomoxetine, or intolerable side effects to atomoxetine

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2008-09; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) Mon-Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milton, Queensland, Australia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zona Centro, Mexico
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fife, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sheffield, South Yorkshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, West Midlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northampton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Period II was a 10-week treatment period. Study Period III was a 4-week period, during which participants continued on atomoxetine treatment in the same dose as given at the end of Study Period II or in a higher dose, up to a maximum of 1.8 mg/kg/day.
Groups:
- Slow Switching Group: Switch from full stimulant dose to atomoxetine 1.2 milligrams per kilogram per day (mg/kg/day), orally (PO), during 10 weeks then continue treatment up to 1.8mg/kg/day, PO to 14 weeks.
- Fast Switching Group: Switch from full stimulant dose to atomoxetine 1.2mg/kg/day, PO, during 2 weeks. Continue atomoxetine 1.2 mg/kg/day to 10 weeks, followed by atomoxetine up to 1.8 mg/kg/day to 14 weeks.
Period: Study Period II
Arm/Group | Slow Switching Group | Fast Switching Group
Started | 57 | 55
Received at Least One Dose of Study Drug | 57 | 54
Completed | 44 | 41
Not Completed | 13 | 14
Not completed — Adverse Event | 3 | 4
Not completed — Lack of Efficacy | 0 | 6
Not completed — Parent/Caregiver Decision | 3 | 0
Not completed — Protocol Violation | 6 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — No drug administered | 0 | 1
Period: Study Period III
Arm/Group | Slow Switching Group | Fast Switching Group
Started | 44 | 41
Completed | 41 | 38
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Parent/Caregiver Decision | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Slow Switching Group: Switch from full stimulant dose to atomoxetine 1.2mg/kg/day, PO, during 10 weeks then continue treatment up to 1.8mg/kg/day, PO to 14 weeks.
- Total: Total of all reporting groups
Arm/Group | Slow Switching Group | Fast Switching Group | Total
Number analyzed (Participants) | 57 | 54 | 111
Age Continuous [Mean (Standard Deviation); unit: years] | 11.1 (2.51) | 12.0 (2.16) | 11.5 (2.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 49 | 44 | 93
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 46 | 43 | 89
  African | 1 | 0 | 1
  Hispanic | 10 | 11 | 21
Region of Enrollment [Number; unit: participants]
  Mexico | 10 | 10 | 20
  Australia | 7 | 5 | 12
  United Kingdom | 8 | 7 | 15
  Spain | 29 | 28 | 57
  Portugal | 3 | 4 | 7
Attention Deficit Hyperactivity Disorder (ADHD) subtype [Number; unit: participants] — ADHD subtype was classified by Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria.
  participants
    Combined | 38 | 36 | 74
    Hyperactive/Impulsive | 1 | 3 | 4
    Inattentive | 17 | 15 | 32
    Not otherwise categorized | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder-Rating Scale (ADHD-RS-IV) Parent Version: Investigator Administered and Scored - Total Score at Week 10 Endpoint
Description: Measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of Attention-Deficit/Hyperactivity Disorder (ADHD). Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54. Higher score indicates greater severity of disease. Least squares means are adjusted for baseline, site, treatment, visit and treatment by visit interaction.
Time Frame: Baseline, 10 weeks
Population: Intention to treat (ITT) population includes all randomized participants who received at least 1 dose of study drug, that is, they have a non-missing dose for atomoxetine study treatment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Slow Switching Group | Fast Switching Group
Number analyzed (Participants) | 57 | 54
units on a scale | -14.3 (1.2) | -15.0 (1.2)
Statistical Analysis 1: Comparison: Slow Switching Group vs Fast Switching Group; Test type: Superiority or Other; p = 0.692, Mixed Models Analysis; Least square mean differences at week 10 = -0.7, 95% CI 2-sided [-4.0 to 2.6], Standard Error of Mean 1.7

2. Secondary Outcome: Change From Baseline in Global Impression of Perceived Difficulties (GIPD) Rating Scale - Patient Total Score at Week 10 Endpoint
Description: The GIPD scale is a 5-item rating of ADHD-related difficulties (overall difficulties perceived in the morning, during school, during homework, in the evening, and over the entire day and night). For each item, difficulties during the past week are rated on a 7-point scale (1 = normal, not difficult at all; 7 = extremely difficult) and the mean of the 5 items is reported. Least square means are adjusted for baseline, site, treatment, visit and treatment by visit interaction.
Time Frame: Baseline, 10 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Slow Switching Group | Fast Switching Group
Number analyzed (Participants) | 57 | 54
units on a scale | -0.6 (0.2) | -0.4 (0.2)
Statistical Analysis 1: Comparison: Slow Switching Group vs Fast Switching Group; Test type: Superiority or Other; p = 0.456, Mixed Models Analysis; Least square mean differences at week 10 = 0.2, 95% CI 2-sided [-0.3 to 0.7], Standard Error of Mean 0.2

3. Secondary Outcome: Change From Baseline in Global Impression of Perceived Difficulties (GIPD) Rating Scale- Parent Total Score at Week 10 Endpoint
Description: as for outcome 2
Time Frame: Baseline, 10 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Slow Switching Group | Fast Switching Group
Number analyzed (Participants) | 57 | 54
units on a scale | -1.0 (0.2) | -0.8 (0.2)
Statistical Analysis 1: Comparison: Slow Switching Group vs Fast Switching Group; Test type: Superiority or Other; p = 0.517, Mixed Models Analysis; Least square mean differences at week 10 = 0.2, 95% CI 2-sided [-0.3 to 0.7], Standard Error of Mean 0.3

4. Secondary Outcome: Change From Baseline in Global Impression of Perceived Difficulties (GIPD) Rating Scale- Investigator Total Score at Week 10 Endpoint
Description: as for outcome 2
Time Frame: Baseline, 10 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Slow Switching Group | Fast Switching Group
Number analyzed (Participants) | 57 | 54
units on a scale | -1.3 (0.2) | -1.2 (0.2)
Statistical Analysis 1: Comparison: Slow Switching Group vs Fast Switching Group; Test type: Superiority or Other; p = 0.526, Mixed Models Analysis; Least square mean differences at week 10 = 0.1, 95% CI 2-sided [-0.3 to 0.6], Standard Error of Mean 0.2

5. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity (CGI-S) Rating Scale - Total Score at Week 10 Endpoint
Description: The CGI- S is a single-item clinician rating of the severity of the participant's ADHD symptoms in relation to the clinician's total experience of ADHD participants. Severity is rated on a seven-point scale (1 = normal, not ill at all; 7 = among the most extremely ill patients). Least square means are adjusted for baseline, site, treatment, visit and treatment by visit interaction.
Time Frame: Baseline, 10 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Slow Switching Group | Fast Switching Group
Number analyzed (Participants) | 57 | 54
units on a scale | -1.7 (0.2) | -1.7 (0.2)
Statistical Analysis 1: Comparison: Slow Switching Group vs Fast Switching Group; Test type: Superiority or Other; p = 0.898, Mixed Models Analysis; Least square mean differences at week 10 = 0.0, 95% CI 2-sided [-0.4 to 0.4], Standard Error of Mean 0.2

6. Secondary Outcome: Change From Baseline in Child Health and Illness Profile Child Edition-Parent Report Form (CHIP-CE-PRF) - Domain Scores at Week 10 Endpoint
Description: CHIP-CE-PRF consists of 76 items. The majority of items assess frequency of activities or feelings using a five-point response format. Standard scores (t-value) were established, with all domains and subdomains having a mean score of 50 and standard deviation (SD) of 10. Standard scores are expressed in SD units. T-score=[(Score- Mean for the reference population [Ref Pop])*10/SD for the Ref Pop]+50. Higher scores mean better quality of life. Least square means are adjusted for baseline, site, treatment, visit and treatment by visit interaction.
Time Frame: Baseline, 10 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: standard deviation units
Arm/Group | Slow Switching Group | Fast Switching Group
Number analyzed (Participants) | 57 | 54
standard deviation units
  Satisfaction Domain | 3.4 (1.6) | 2.2 (1.6)
  Comfort Domain | 0.7 (1.2) | 4.1 (1.1)
  Risk Avoidance Domain | 4.9 (1.4) | 2.9 (1.4)
  Resilience Domain | 1.8 (1.4) | -1.0 (1.4)
  Achievement Domain | 3.5 (1.7) | -1.2 (1.6)

7. Secondary Outcome: Change From Baseline in Treatment Satisfaction Preference Survey Mean Score at Week 10 Endpoint
Description: The Treatment Satisfaction Survey consists of a five-question survey each rated on a 5 point scale (0=very satisfied/very likely, 4=very dissatisfied/not at all likely). The mean score over the items is reported.
Time Frame: Baseline, 10 weeks
Population: Intention to treat (ITT) population includes all randomized participants who received at least 1 dose of study drug, that is, they have a non-missing dose for atomoxetine study treatment. Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Slow Switching Group | Fast Switching Group
Number analyzed (Participants) | 53 | 53
units on a scale | -0.7 (1.16) | -0.5 (1.11)

8. Secondary Outcome: Change From Baseline in Blood Pressure (BP) at Week 6 and Week 14 Endpoint
Time Frame: Baseline, 6 weeks, 14 weeks
Population: Intention to treat (ITT) population includes all randomized participants who received at least 1 dose of study drug, that is, they have a non-missing dose for atomoxetine study treatment, and with both baseline and week 6 or 14 values.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Slow Switching Group | Fast Switching Group
Number analyzed (Participants) | 57 | 54
mmHg
  Week 6 Change Diastolic BP (n=52, 52) | 1.5 (7.21) | 1.9 (8.31)
  Week 6 Change Systolic BP (n=52, 52) | 1.2 (7.74) | 0.5 (9.05)
  Week 14 Change Diastolic BP (n=43, 40) | 2.3 (7.58) | 3.1 (7.04)
  Week 14 Change Systolic BP (n= 43, 40) | -0.2 (8.62) | 2.6 (9.00)

9. Secondary Outcome: Change From Baseline in Pulse Rate at Week 6 and Week 14 Endpoint
Time Frame: Baseline, 6 weeks, 14 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Slow Switching Group | Fast Switching Group
Number analyzed (Participants) | 57 | 54
beats per minute
  Week 6 Change (n=52, 52) | 6.8 (11.12) | 4.2 (8.83)
  Week 14 Change (n=43, 40) | 3.4 (12.69) | 5.9 (10.17)

10. Primary Outcome: Change From Baseline in ADHD-RS-IV Parent Version: Investigator Administered and Scored - Total Score at Week 2 Endpoint
Description: Measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of ADHD. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54. Higher score indicates greater severity of disease. Least squares means are adjusted for baseline, site, treatment, visit and treatment by visit interaction.
Time Frame: Baseline, 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Slow Switching Group | Fast Switching Group
Number analyzed (Participants) | 57 | 54
units on a scale | -8.0 (1.0) | -8.1 (1.0)
Statistical Analysis 1: Comparison: Slow Switching Group vs Fast Switching Group; Test type: Superiority or Other; p = 0.927, Mixed Models Analysis; Least square mean differences at week 2 = -0.1, 95% CI 2-sided [-2.9 to 2.6], Standard Error of Mean 1.4

11. Secondary Outcome: Change From Baseline in Body Weight at Week 6 and Week 14 Endpoint
Time Frame: Baseline, 6 weeks, 14 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Slow Switching Group | Fast Switching Group
Number analyzed (Participants) | 57 | 54
kilogram
  Week 6 Change (n=52, 52) | -0.4 (1.12) | 0.6 (1.25)
  Week 14 Change (n=43, 40) | 0.6 (1.64) | 1.1 (2.15)

12. Secondary Outcome: Number of Participants With Suicidal Behaviors and Ideations
Description: Columbia Suicide Rating Scale (C-SSRS): scale capturing occurrence, severity, and frequency of suicide-related thoughts and behaviors. Number of participants with suicidal behaviors and ideations are provided. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions, which includes wish to be dead, and 4 different categories of active suicidal ideation.
Time Frame: Baseline through 14 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Slow Switching Group | Fast Switching Group
Number analyzed (Participants) | 57 | 54
participants | 1 | 1

ADVERSE EVENTS:
Arm/Group | Slow Switching Group | Fast Switching Group
Serious Adverse Events (participants affected / at risk) | 1/57 | 1/54
Other Adverse Events (participants affected / at risk) | 35/57 | 30/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Slow Switching Group (N=57) | Fast Switching Group (N=54)
VIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Slow Switching Group (N=57) | Fast Switching Group (N=54)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 6 (13)
Abdominal pain upper (Gastrointestinal disorders) | 8 (11) | 5 (5)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (6)
Fatigue (General disorders) | 3 (3) | 4 (4)
Irritability (General disorders) | 4 (5) | 3 (3)
Pyrexia (General disorders) | 4 (4) | 2 (3)
Nasopharyngitis (Infections and infestations) | 7 (8) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 11 (12) | 7 (7)
Headache (Nervous system disorders) | 11 (16) | 12 (19)
Somnolence (Nervous system disorders) | 4 (4) | 9 (9)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days